CLINICAL TRIAL: NCT04473625
Title: Stool Collection Sub-Study of Exact Sciences Protocol 2018-01: "Blood Sample Collection to Evaluate Biomarkers in Subjects With Untreated Solid Tumors
Brief Title: Stool Collection Sub-Study of Exact Sciences Protocol 2018-01
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-01B
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer; Colo-rectal Cancer; Cancer
Keywords: Colorectal Cancer; Cologuard; Sample Collection
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool Collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Breast: Subjects with clinically confirmed breast cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Lung: Subjects with clinically confirmed lung cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Colorectal: Subjects with clinically confirmed colorectal cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Prostate: Subjects with clinically confirmed prostate cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Bladder: Subjects with clinically confirmed or suspicion of bladder cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Uterine: Subjects with clinically confirmed uterine cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Kidney/Renal Pelvis: Subjects with clinically confirmed or suspicion of kidney/renal pelvis cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Ovarian: Subjects with clinically confirmed or suspicion of ovarian cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Liver: Subjects with clinically confirmed liver cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Pancreas: Subjects with clinically confirmed or suspicion of pancreatic cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Stomach: Subjects with clinically confirmed stomach cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection
- Esophageal: Subjects with clinically confirmed esophageal cancer and who are treatment naive will provide a stool sample within 30 days of enrollment. No additional stool sample collections will occur.
  Interventions: Other: Stool Sample Collection

INTERVENTIONS:
Other: Stool Sample Collection — Subjects participating in the study will provide a stool sample within 30 days of enrollment.

SUMMARY:
The primary objective of this sub-study is to obtain de-identified, clinically characterized, stool specimens from subjects with untreated solid tumors for research use in the development and validation of a stool-based test for colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is currently enrolled in Exact Sciences Protocol 2018-01.
* Subject is willing and able to provide a stool sample.
* Subject understands the study procedures and is able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the sub-study protocol, or put the person at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women, 18 years of age or older, who enroll in Exact Sciences Protocol 2018-01. Approximately 450 subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Stool-based test for colorectal cancer | Point in time (one day) stool collection within 30 days of enrollment
  Research for the development and validation of a stool-based test for colorectal cancer

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Marin Cancer Care, Greenbrae, California
  - Easter Ct Hematology, Norwich, Connecticut
  - CSNF- Central Business Office, Jacksonville, Florida
  - Park Nicollet Institute - Oncology Research, Saint Louis Park, Minnesota
  - St. Dominic's Gynecologic Oncology, Jackson, Mississippi
  - Cone Health Cancer Center, Greensboro, North Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Community Cancer Trials of Utah, Ogden, Utah
  - CAMC Clinical Trials Center, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol and informed consent form (when applicable) will also be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.